CLINICAL TRIAL: NCT04676087
Title: Mogamulizumab and Extracorporeal Photopheresis (ECP) for the Treatment of Sézary Syndrome and Erythrodermic Mycosis Fungoides, a Phase 1b/2 Study
Brief Title: Mogamulizumab and Extracorporeal Photopheresis for the Treatment of Sezary Syndrome or Mycosis Fungoides
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela Allen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001265; NCI-2020-06013 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP5101-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-11-09; First posted 2020-12-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Mycosis Fungoides; Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Sezary Syndrome
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Sezary Syndrome | interventions — Photopheresis; mogamulizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (mogamulizumab, ECP) (Experimental): INDUCTION (WEEKS 1-7): Patients receive mogamulizumab IV over 60 minutes on days 1, 8, 15, 22, and 36 in the absence of disease progression progression and unacceptable toxicity. Patients also undergo extracorporeal photopheresis on days 1, 8, 15, 22, 29, and 36 in the absence of disease progression and unacceptable toxicity.
  TREATMENT (CYCLES 1-12): Patients receive mogamulizumab IV over 60 minutes on days 1 and 15, and undergo extracorporeal photopheresis on days 1 and 15 of cycles 1-6, then day 1 of subsequent cycles. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression and unacceptable toxicity.
  MAINTENANCE (CYCLES 13+): Patients with clinical benefit may continue extracorporeal photopheresis on day 1. Cycles repeat every 28 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Procedure: Extracorporeal Photopheresis; Biological: Mogamulizumab; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis — Undergo ECP
  Other Names: Extracorporeal Photophoresis; photopheresis; Photophoresis
Biological: Mogamulizumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(CC Chemokine Receptor CCR4) (Human-Mouse Monoclonal KW-0761 Heavy Chain), Disulfide With Human-Mouse Monoclonal KW-0761 Kappa-Chain, Dimer; KM8761; KW-0761; Mogamulizumab-kpkc; Poteligeo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase Ib/II trial investigates the side effects of mogamulizumab and extracorporeal photopheresis and to see how well they work in treating patients with Sezary syndrome or mycosis fungoides. Mogamulizumab (a humanized antibody) binds to CCR4, a protein often found in high amounts on T-cell lymphoma cells. Binding to these cells may slow their growth, as well as mark them for attack by the immune system. Extracorporeal photopheresis (ECP) is a standard treatment for cancers that affects the skin, and may work by killing some lymphoma cells directly and by boosting the body's immune response against other lymphoma cells. Giving mogamulizumab together with ECP may work better in treating patients with Sezary syndrome or mycosis fungoides compared to either therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of mogamulizumab and ECP in Sezary syndrome (SS) and erythrodermic mycosis fungoides (MF).

II. To determine the efficacy of the combination of mogamulizumab and extra-corporeal photopheresis in SS and erythrodermic MF.

SECONDARY OBJECTIVE:

I. To assess response by disease compartment, time to response, duration of response, progression free survival (PFS), and change in quality of life in patients with Sezary syndrome and erythrodermic MF treated with mogamulizumab and ECP.

TERTIARY/EXPLORATORY OBJECTIVE:

I. To assess biomarkers of response and changes in immunologic response on serial blood samples and peripheral blood flow cytometry.

OUTLINE:

INDUCTION (WEEKS 1-7): Patients receive mogamulizumab intravenously (IV) over 60 minutes on days 1, 8, 15, 22, and 36 in the absence of disease progression progression and unacceptable toxicity. Patients also undergo extracorporeal photopheresis on days 1, 8, 15, 22, 29, and 36 in the absence of disease progression and unacceptable toxicity.

TREATMENT (CYCLES 1-12): Patients receive mogamulizumab IV over 60 minutes on days 1 and 15, and undergo extracorporeal photopheresis on days 1 and 15 of cycles 1-6, then day 1 of subsequent cycles. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression and unacceptable toxicity.

MAINTENANCE (CYCLES 13+): Patients with clinical benefit may continue extracorporeal photopheresis on day 1. Cycles repeat every 28 days in the absence of disease progression and unacceptable toxicity.

After completion of study treatment, patients are followed up for 90 days, then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Histopathologic diagnosis of primary cutaneous T-cell non-Hodgkin lymphoma (CTCL) (mycosis fungoides [MF] or Sezary syndrome [SS]), confirmed by skin biopsy, or lymph node, or blood assessment, of current disease
* CTCL stage 3A-4A2 disease at study entry according to International Society of Cutaneous Lymphoma (ISCL)/European Organization for Research and Treatment of Cancer (EORTC)
* Newly diagnosed or =< 3 different lines of systemic therapy

  * Systemic therapy includes oral retinoids, interferon, pralatrexate, methotrexate, vorinostat, romidepsin, single or multi-agent chemotherapy or other oral, IV or subcutaneous treatments used to treat systemic disease
  * A line of therapy is defined as any therapy or group of therapies that was started or changed for lack of response, disease progression, or intolerance
* Prior cytotoxic chemotherapy excluding low dose methotrexate
* A minimum washout period of 4 weeks after previous CTCL therapy is recommended prior to the first dose of combination therapy
* Willing and able to comply with all aspects of the protocol
* Provide voluntary written informed consent prior to any study specific screening procedures
* Absolute neutrophil count (ANC) >= 500/mcL (within 16 days of cycle 1 day 1)
* Platelets >= 50,000/mcL (within 16 days of cycle 1 day 1)
* Total bilirubin =< 3 institutional upper limit of normal (ULN) (within 16 days of cycle 1 day 1)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5 institutional upper limit of normal (ULN) (within 16 days of cycle 1 day 1)
* Not dialysis dependent, creatinine clearance >= 30 mL/min (within 16 days of cycle 1 day 1)
* Female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy: documented by negative beta-human chorionic gonadotropin [beta-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of beta-hCG. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
* FCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 30 Days after completion. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 30 days after completion of study drug administration. A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months

Exclusion Criteria:

* Visceral involvement except for CTCL involvement of the bone marrow
* Bulky lymphadenopathy (> 5 cm), or pathologically N3 lymph node involvement
* Total skin electron beam therapy within 6 months prior to registration
* Prior allogeneic transplantation
* Prior mogamulizumab therapy within 6 months of registration or progression or intolerance of mogamulizumab
* Patients with 2 or less doses of prior mogamulizumab prior to registration will be eligible regardless of date mogamulizumab was received

  * Patients who received mogamulizumab pre-study enrollment would restart day 1 dosing per protocol
* Prior ECP > 2 months in duration within 3 months of registration
* Patients with ECP treatment prior to registration will be eligible regardless of date ECP was received (as long as it was not > 2 months in duration within the 3 months immediately prior to registration), as long as they have measurable disease at the time of enrollment
* Use of topical steroids within 14 days of day 1 of initial therapy is not allowed, with the following exception:

  * Topical steroids or systemic low dose steroids (=< 10 mg/day prednisone) are allowed in subjects with erythroderma who have been on corticosteroids for a prolonged period of time and where discontinuation may lead to rebound flare in disease. The concomitant steroid medication is allowed as long as the type of steroid, route of administration, and steroid dose remain the same as what the subject had been receiving for a prolonged period of time
* Severe or uncontrolled autoimmune condition
* Active, life threatening malignancy (except for CTCL, definitively treated basal or squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix, or other localized malignancies treated with curative intent with surgery or radiation alone) within the past 12 months
* Serious intercurrent illness
* Known significant cardiac disease requiring ongoing treatment, including congestive heart failure (CHF), severe coronary artery disease (CAD), cardiomyopathy, uncontrolled cardiac arrhythmia, unstable angina pectoris, or myocardial infarction (MI) (within 6 months of study enrollment)
* Major surgery within 2 weeks of study enrollment
* Significant or uncontrolled infections requiring systemic anti-infective therapy
* Patients with human immunodeficiency virus (HIV) infection are eligible. Patients with HIV infection must meet the following: No evidence of co-infection with hepatitis B or C; CD4+ count > 400/mm; no evidence of resistant strains of HIV; on anti-HIV therapy with an HIV viral load < 50 copies HIV RNA/mL. Patients with HIV must have ongoing follow-up with an infectious disease specialist and must have been evaluated within 90 days of cycle 1 day 1
* Patients with a history of hepatitis C are eligible as long as the hepatitis C has been treated and cleared and they have no evidence of hepatic dysfunction related to hepatitis C. Patients must have been seen by a hepatologist within 6 months of cycle 1 day 1
* Patients who test positive for hepatitis B core antibody may enroll on the study as long as they test negative for both hepatitis B surface antigen and hepatitis B deoxyribonucleic acid (DNA), and if they have no evidence of hepatic dysfunction that is felt to be related to hepatitis B
* Patients may not have an auto-immune disease requiring systemic immunosuppression, biologic therapy, and/or steroid use (>= 10 mg daily of prednisone or equivalent)
* Patients will not be excluded based on CCR4 expression
* Females who are pregnant (positive urine test) or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (DLT's) (Phase Ib) | Up to 6 weeks
  Descriptive statistics (n, frequency and percentage) of toxicities and number of DLT's during the DLT window per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported. Corresponding listings of data will be generated. DLT rate will be calculated as proportion (Patients with DLT/Total patients) along with 95% confidence intervals using the Clopper-Pearson method.
Rate of overall response lasting at least 6 months (ORR6) (Phase II) | Up to 3 years post treatment
  Assessed using the Global Response Score (GRS). ORR6 rate will be determined by dividing the number of ORR6's by the total number of evaluable patients. Will be calculated as proportion (Responders/Total patients) along with 95% confidence intervals using the Clopper-Pearson method. Chi-square test or Fisher's exact test will be used to compare the efficacy in term of response rate between the different groups stratified by baseline factors, respectively. Logistic regression model will be further employed to test the adjusted effect of dosage on the response rate after adjusting for other clinical factors and demographic factors.

SECONDARY OUTCOMES:
Best overall response rate (ORR) | Up to 3 years post treatment
  Assessed using the Global Response Score (GRS), which consists of skin evaluation (modified severity weighted assessment tool [mSWAT]), radiographic assessment, and detection of circulating Sezary cells on flow cytometry in patients that have received at least 1 month of combined therapy. Overall response, complete response, and partial response will be calculated as proportions along with 95% confidence intervals using the Clopper-Pearson method.
Duration of response (DOR) | Up to 3 years post treatment
  Based on GRS. Defined as time from the date when criteria for response (complete response [CR] or partial response [PR]) based on GRS was first met until the date when the response was first lost (date of loss is date when first meets criteria for progressive disease [PD] or death). Will be estimated using the Kaplan-Meier method.
Time to response (TTR) | Up to 3 years post treatment
  Based on GRS. Defined as time from the date of first dosing to the date when criteria for response (CR or PR) based on GRS are first met. Will be estimated using the Kaplan-Meier method.
Overall survival (OS) | Date of 1st dose of study drug to death from any cause, assessed up to 3 years
  Estimated by Kaplan-Meier method. Cox proportional hazards models will be further used in the multivariable analyses to assess the patients' OS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.
Progression free survival (PFS) | Date of 1st dose of study drug to progression, death, or subsequent systemic anti-cancer therapy, assessed up to 3 years
  Estimated by Kaplan-Meier method. Cox proportional hazards models will be further used in the multivariable analyses to assess the patients' PFS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.
Incidence of adverse events | Up to 3 years post treatment
  Adverse events (AEs) will be listed and summarized. Adverse events will also be listed by severity, seriousness, and by system organ class. Will also evaluate toxicities which will be presented in tabular form as appropriate based on grade and attribution. The number and percentage of subjects who experience AEs will be presented in tabular and/or graphical format and summarized descriptively, where appropriate AEs will be presented with and without regard to causality based on the investigator's judgment. The frequency of overall toxicity, categorized by toxicity grades 1 through 5, will be described. Additional summaries will be provided for AEs that are observed with higher frequency.

OTHER OUTCOMES:
Genomic and immunologic profiles | Up to 3 years post treatment
  Correlation of baseline genomic and immunologic profiles with response. Will analyze baseline samples using hierarchical clustering to identify patterns associated with different response patterns and kinetics. Will describe baseline immunologic profiles descriptively.
T cell populations will include T-regulatory cells and CD8+ cytotoxic T-cells | Induction is 7 weeks. Treatment consists of 28 cycles (12). Maintenance resumes after 12 cycles with ECP on day 1 of each 28 day cycle.
  Cytokines will be assessed via the Luminex panel.
Changes in genomic profiles | Induction is 7 weeks. Treatment consists of 28 cycles (12). Maintenance resumes after 12 cycles with ECP on day 1 of each 28 day cycle.
  Measuring genomic profiles of the tumor and immune cells from peripheral blood and biopsy samples at specific time points.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela B Allen, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States